CLINICAL TRIAL: NCT07332637
Title: Evaluation of the Relationship Between 0-24-Hour Fraction of Inspired Oxygen (FiO₂) Exposure and Changes in the Uric Acid/Albumin Ratio in Intensive Care Unit Patients Diagnosed With Sepsis
Brief Title: Association Between Early FiO₂ Exposure and Changes in the Uric Acid/Albumin Ratio in Septic ICU Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assos.Prof., Istinye University
Other Study IDs: 329-2025
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Hyperoxia / High FiO₂ Exposure; Uric Acid/Albumin Ratio (UAR)
MeSH Terms: conditions — Hyperoxia | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Oxygen Exposure (Fraction of Inspired Oxygen, FiO₂) - Standard of Care (Observational, No Experimental Intervention) — This study does not involve an experimental intervention. Patients will receive oxygen therapy as part of standard clinical care according to routine intensive care unit protocols and clinical indications. Fraction of inspired oxygen (FiO₂) levels administered during the first 24 hours of ICU admission will be recorded from ventilator and oxygen delivery system data. No changes will be made to patients' diagnostic, therapeutic, or oxygen administration practices. The study is purely observational, and collected data will be used to evaluate the association between FiO₂ exposure and changes in the uric acid/albumin ratio.

SUMMARY:
This prospective, non-interventional study aims to investigate the relationship between early oxygen exposure and oxidative stress in adult intensive care unit (ICU) patients diagnosed with sepsis or septic shock. Fraction of inspired oxygen (FiO₂) levels administered during the first 24 hours of ICU admission will be evaluated in relation to changes in the uric acid/albumin ratio (UAR), a biochemical marker reflecting oxidative burden and inflammation. Serum uric acid and albumin levels will be measured at ICU admission and at 24 hours, and the percentage change in UAR (ΔUAR%) will be calculated. Associations between FiO₂ exposure parameters and ΔUAR% will be analyzed, along with secondary outcomes including 28-day mortality and oxygenation indices. The findings may help clarify whether excessive oxygen therapy contributes to oxidative stress and whether UAR can serve as an accessible biomarker of oxygen-related oxidative injury in septic ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older
* Admission to the intensive care unit with a diagnosis of sepsis according to Sepsis-3 criteria
* Receipt of oxygen therapy with FiO₂ ≥ 0.3 during ICU stay
* Availability of serum uric acid, albumin, and lactate measurements and calculated SOFA scores at ICU admission
* Availability of serum uric acid and albumin levels both at ICU admission (baseline) and at 24 hours
* Provision of informed consent by the patient or a legally authorized representative

Exclusion Criteria:

* Age younger than 18 years
* Pregnant or breastfeeding women
* Chronic kidney disease or receipt of renal replacement therapy
* Advanced liver failure (Child-Pugh class C)
* Receipt of albumin infusion within the previous 24 hours
* Use of medications that affect uric acid metabolism (e.g., allopurinol, febuxostat, rasburicase)
* History of active gout attack or malignancy-related hyperuricemia
* Missing serum uric acid or albumin measurements at baseline or 24 hours
* Inability to obtain informed consent from the patient or a legally authorized representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years and older who are admitted to a tertiary-level intensive care unit with a diagnosis of sepsis or septic shock according to Sepsis-3 criteria. All included patients receive oxygen therapy as part of standard clinical care, with a fraction of inspired oxygen (FiO₂) of at least 0.3 during the early phase of ICU admission. The population represents critically ill patients requiring close monitoring, respiratory support, and comprehensive laboratory evaluation. Patients with conditions or treatments that may independently affect uric acid or albumin metabolism are excluded to allow a clearer assessment of the relationship between oxygen exposure and changes in the uric acid/albumin ratio.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Uric Acid/Albumin Ratio in Relation to Early FiO₂ Exposure | From ICU admission (0 hour) to 24 hours after admission
  The primary outcome is the association between fraction of inspired oxygen (FiO₂) levels administered during the first 24 hours of intensive care unit admission and the change in the uric acid/albumin ratio (UAR). Serum uric acid and albumin levels will be measured at ICU admission (baseline) and at 24 hours, and the percentage change in UAR (ΔUAR%) will be calculated. Correlation analyses will be performed to evaluate the relationship between FiO₂ exposure parameters and ΔUAR%

REFERENCES:
- [Background] Katakam SN, Cherukuri M, Kada M, Hanji P, Kudru CU. The Prognostic Significance of Serum Uric Acid in Sepsis: A Comparative Study on Adult Patients. Indian J Crit Care Med. 2025 May;29(5):407-412. doi: 10.5005/jp-journals-10071-24968. Epub 2025 May 8. PMID 40416537
- [Background] Ertan OES, Gokce O, Bal C, Kocaturk E, Ertan O, Mutluay R. Investigation of the Relationship Between Serum Uric Acid-to-Albumin Ratio and 28-Day Mortality in Patients With and Without Acute Kidney Injury. J Acute Med. 2024 Dec 1;14(4):152-159. doi: 10.6705/j.jacme.202412_14(4).0003. PMID 39624148